CLINICAL TRIAL: NCT06882044
Title: The Effect of a Mobile Application on Treatment Adherence, Self-Management, and Quality of Life in Patients With Acute Myocardial Infarction Undergoing Primary Percutaneous Coronary Intervention
Brief Title: The Effect of a Mobile Application in Patients With Acute Myocardial Infarction
Acronym: Mobileapp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Trakya University (Other)
Responsible Party: Principal Investigator, Ezgi Kınıcı Dirik, Principal Investigator, Trakya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TÜTF-BAEK 2021/283; There is no funding support (Other: There is no funding support for the study)
Record Dates: First submitted 2025-02-06; First posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Acute Myocardial Infarction (AMI); Mobile Health Technology (mHealth); Quality of Lifte; Treatment Adherence; Self Care
Keywords: Mobile health application; acute myocardial infarction; treatment adherence; self-care management; quality of life
MeSH Terms: conditions — Treatment Adherence and Compliance

STUDY DESIGN:
Intervention Model Description: Prospective (6-month follow-up), two-group (control and intervention), randomised controlled, experimental study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Group receiving standard discharge education with 'Educational Booklet for Patients Who Have Had a Heart Attack'
- Intervention group (Experimental): Group receiving standard discharge education with 'Educational Booklet for Patients Who Have Had a Heart Attack' and using Mobile Health Application (mHealth)
  Interventions: Device: mHealth

INTERVENTIONS:
Device: mHealth — The mobile application contains medication and personalised reminders, the screen where blood pressure and pulse are entered, the lifestyle change recommendations information, and the section that allows users to communicate with the researcher. Also, there is a control panel that allows the application to be controlled remotely, patient information to be viewed, data to be monitored, lifestyle information to be uploaded and viewed in the mHealth, personalised reminders to be sent to patients, and communication with patients.
  Arms: Intervention group

SUMMARY:
Background and Aim: Acute myocardial infarction is a clinical condition with high mortality and morbidity rates. Ensuring patient adherence to treatments and lifestyle recommendations after discharge is crucial for effective post-acute myocardial infarction management. This study aimed to determine the impact of a mobile application on treatment adherence, self-management, and quality of life in patients with acute myocardial infarction undergoing primary percutaneous coronary ıntervention.

Material and Methods: This randomized controlled and experimental study was conducted between 2021 and 2024 at the cardiology clinic of a university hospital. It included patients who had their first time with ST-segment elevation acute myocardial infarction and underwent primary percutaneous coronary intervention (n=31/30).

The control group was provided standard discharge education with the "Educational Booklet for Patients Who Have Had a Heart Attack". The intervention group, in addition to these practices, mobile application support was provided. They were followed up for 6 months post-discharge. Data were collected at 1, 3 and 6 months. The patient information form including characteristics related to lifestyle changes, Medication Adherence Reporting Scale (MARS), and Myocardial Infarction Dimensional Assessment Scale (MIDAS) were used in data collection.

DETAILED DESCRIPTION:
Aim of the study The aim of this study was to determine the effect of the mHealth on treatment adherence, and quality of life in patients with acute myocardial infarction undergoing Primary Percutaneous Coronary Intervention (PPCI).

Methods The study was a prospective (6-month follow-up), two-group (control and intervention), randomised controlled, experimental study, between 2021 and 2024.

The universe of the study consisted of patients who had their first time ST Segment Elevation Myocardial Infarction (STEMI) undergoing PPCI in the Cardiology Clinic of a university hospital in western Turkey. In determining the sample of the study, power analysis was performed with reference to the study of Turan Kavradım and Özer. The effect size of the study was found to be 0.92. Based on this effect size, it was determined that it was sufficient to include a total of 54 patients, 27 in each group, at 95% power and 0.05 significance level. However, considering a 20% loss rate during the study period, it was aimed to reach a total of 66 patients, 33 patients for each group (30). The selection of patients to the intervention and control groups was made using the simple randomization method. According to the randomization list, the groups were matched based on the time of discharge from the clinic of the patients. For patients who were discharged on the same day, the matching was based on their hospitalization times. The inclusion criteria were as follows: the patients who (i) had first time STEMI undergoing PPCI, (ii) are over 18 years of age, (iii) have a smartphone, (iv) have internet access, (v) have orientation to place, time and situation, (vi) have no problems with vision, hearing and speech, (vii) are at least literate, (viii) regularly come in for the doctor's check up, and (ix) volunteer to participate in the study. Among the volunteers participating in the study, those who wanted to leave the study (2 patients) and those who

didn't come in for the doctor's check up (3 patients) were excluded from the follow-up. Therefore, the study was completed with 61 patients, 30 in the intervention group and 31 in the control group. CONSORT flow diagram of the phases of the study is displayed in Figure 1.

Study Protocol

In the study, the control group was given a standard discharge education with an educational booklet. The intervention group was provided mHealth support, in addition to that practice. Within the scope of standard discharge education, firstly an educational booklet was developed, and this booklet was given to all patients.

Educational booklet

It was created to provide self-management in patients with AMI. During the development phase of the educational booklet, expert opinions were obtained from a total of 9 people, including 3 cardiologists, 4 academic nurses and 2 cardiology nurses, and the final version of it was created.

mHealth and web page control panel

Firstly, the content of the application was determined based on the education booklet and sample mHealth studies in the literature. In order to evaluate the content of the mHealth, expert opinions were obtained from 3 cardiologists, 4 academic nurses and 2 cardiology nurses. Then, a software company was contacted and the mHealth called "MEDIFOLL" was developed. The interface of the application includes "Medication Information", Blood P. & Pulse", 'Notifications', 'Lifestyle' and 'Contact' sections. In the "Medication Information" section, medication entries are made. When it is time to take each medication, the mHealth sends a medication reminder notification to the user. "Blood P. & Pulse" section includes the screen where blood pressure and pulse are entered. The "Notifications" section displays personalized reminders sent by the researcher to the users via the web page control panel. Personalized reminders are information regarding LCR which are included in the education booklet. The "Lifestyle" section contains the information contained in the booklet regarding LCR. The "Contact" section allows users to communicate with the researcher. In this way, patients can send their questions to the researcher via message. After mHealth was developed, a web page control panel was created that allows the mHealth to be controlled remotely, patient information to be viewed, data to be monitored, lifestyle information to be uploaded and

viewed in the mHealth, personalized reminders to be sent to patients, and to be communicated with patients. Additionally, the application was uploaded the Google Play Store and App Store. The mHealth and website were tested by experts for 1 week to determine usability of them and errors. Finally, a pilot study was conducted with 4 patients and the patients were allowed to use the application for a month. Patients who participated in the pilot study were not included in the study.

After the pilot study was completed, the Patient Information Form was filled out with all patients in the patient room before discharge. The researcher provided training to the patients in both groups in line with the educaiton booklet and it was delivered to the patients. MEDIFOLL application was downloaded to the mobile phones of the patients in the intervention group and user registration was made. Information was provided to them on how to use the application and how to enter data such as blood pressure and pulse rate. The times of the use of medications prescribed during discharge were planned together with the patients and they were provided with the opportunity to enter their medications into the application. Then, all patients were interviewed in the outpatient clinic at 1, 3, and 6 months following their discharge and The Patient Information Form, MARS, and MIDAS scales were filled out. The flow chart of the research is presented in Figure 2.

Data collection tool

Patient Information Form: It, developed by the researcher through a literature review, consists of questions about the socio-demographic, the lifestyle, and the disease characteristics of the participants.

Medical Adherence Report Scale (MARS): The scale was developed by Horne and Hankins to determine medication adherence in individuals with chronic diseases. The Turkish validity and reliability of the scale was performed by Şen et al. The scale has 5 items, one sub-dimension and 5-point Likert type. The total score obtained from the scale varies between 5 and 25. A high total score indicates adherence to medication treatment, while a low score indicates non-adherence to medication treatment.

Myocardial Infarction Dimensional Assessment Scale (MIDAS): The Turkish validity and reliability of the scale, developed by Thompson et al., was performed by Yılmaz et al. The scale is used to determine the HRQoL of individuals with MI and consists of 35 items and 7 sub-dimensions (physical activity, insecurity, emotional reaction, dependency, diet, concerns over medication, and medication side effects). This 5-point Likert-type scale is scored between 0-4. Scores that can be obtained from the scale and its sub-dimensions vary between 0-100. The score is calculated with the formula: (Total score obtained from the sub-dimension/highest score that can be obtained from the sub-dimension) x100. As the scores obtained from the scale increase, the perceived HRQoL worsens.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had ST-segment elevation acute myocardial infarction and underwent primary percutaneous coronary intervention,
* Above the age of 18,
* Have a smart phone,
* Have internet access,
* Have orientation to place, time, and situation,
* Have no problems with vision, hearing, or speech,
* Have minimal literacy,
* Patients who volunteer to participate in the study

Exclusion Criteria:

* Patients who want to leave the study,
* Patients who do not come to their doctor's check-ups regularly.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-07-10 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
Medication adherence | at 1, 3, and 6 months following their discharge
  Medication Adherence Report Scale: The total score obtained from the scale varies between 5 and 25. A high total score indicates adherence to medication treatment, while a low score indicates non-adherence to medication treatment.
Self-management | at 1, 3, and 6 months following their discharge
  This title contains adherence of individuals to lifestyle change recommendations. The questions in this section are: Status of smoking, status of regular physical activity/exercise (>150 min/week), status of consumption of fruit and vegetables per ≥5 days a week and status of consumption of <500 g of red meat per week.

SECONDARY OUTCOMES:
Quality of life of individuals with Myocardial Infarction | at 1, 3, and 6 months following their discharge
  Myocardial Infarction Dimensional Assessment Scale (MIDAS): The scale is used to determine the quality of life of individuals with Myocardial Infarction. Scores that can be obtained from the scale and its sub-dimensions vary between 0-100. As the scores obtained from the scale increase, the perceived quality of life worsens.

CONTACTS AND LOCATIONS:
Overall Officials: Eylem Paslı Gürdoğan, Ass. Prof., Study Director — Trakya University
Locations (1):
- Trakya University, Edirne, Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harbi AS, Soh KL, Yubbu PB, Soh KG. The impact of cardiac rehabilitation on psychosocial factors, functional capacity, and left ventricular function in patients with coronary artery disease: Systematic review and meta-analysis. F1000Research. 2024;13:575
- [Background] Delgado-Lista J, Alcala-Diaz JF, Torres-Pena JD, Quintana-Navarro GM, Fuentes F, Garcia-Rios A, Ortiz-Morales AM, Gonzalez-Requero AI, Perez-Caballero AI, Yubero-Serrano EM, Rangel-Zuniga OA, Camargo A, Rodriguez-Cantalejo F, Lopez-Segura F, Badimon L, Ordovas JM, Perez-Jimenez F, Perez-Martinez P, Lopez-Miranda J; CORDIOPREV Investigators. Long-term secondary prevention of cardiovascular disease with a Mediterranean diet and a low-fat diet (CORDIOPREV): a randomised controlled trial. Lancet. 2022 May 14;399(10338):1876-1885. doi: 10.1016/S0140-6736(22)00122-2. Epub 2022 May 4. PMID 35525255
- [Background] Berg E, Agewall S, Brolin EB, Caidahl K, Cederlund K, Collste O, Daniel M, Ekenback C, Jensen J, Y-Hassan S, Henareh L, Maret E, Spaak J, Sorensson P, Tornvall P, Lynga P. Health-related quality-of-life up to one year after myocardial infarction with non-obstructive coronary arteries. Eur Heart J Qual Care Clin Outcomes. 2023 Sep 12;9(6):639-644. doi: 10.1093/ehjqcco/qcac072. PMID 36328780
- [Background] Lao SSW, Chair SY, Wang Q, Leong MLT. The Feasibility and Effects of Smartphone-Based Application on Cardiac Rehabilitation for Patients After Percutaneous Coronary Intervention: A Randomized Controlled Trial. J Cardiovasc Nurs. 2024 Jan-Feb 01;39(1):88-101. doi: 10.1097/JCN.0000000000000993. Epub 2023 May 11. PMID 37088896
- [Background] Lizcano-Alvarez A, Carretero-Julian L, Talavera-Saez A, Cristobal-Zarate B, Cid-Exposito MG, Alameda-Cuesta A; REccAP Group (Red de Enfermeria de Cuidados Cardiovasculares en Atencion Primaria). Intensive nurse-led follow-up in primary care to improve self-management and compliance behaviour after myocardial infarction. Nurs Open. 2023 Aug;10(8):5211-5224. doi: 10.1002/nop2.1758. Epub 2023 Apr 21. PMID 37084014
- [Background] Bhagavathula AS, Aldhaleei WA, Atey TM, Assefa S, Tesfaye W. Efficacy of eHealth Technologies on Medication Adherence in Patients With Acute Coronary Syndrome: Systematic Review and Meta-Analysis. JMIR Cardio. 2023 Dec 19;7:e52697. doi: 10.2196/52697. PMID 38113072
- [Background] Krackhardt F, Jornten-Karlsson M, Waliszewski M, Knutsson M, Niklasson A, Appel KF, Degenhardt R, Ghanem A, Kohler T, Ohlow MA, Tschope C, Theres H, Vom Dahl J, Karlson BW, Maier LS. Results from the "Me & My Heart" (eMocial) Study: a Randomized Evaluation of a New Smartphone-Based Support Tool to Increase Therapy Adherence of Patients with Acute Coronary Syndrome. Cardiovasc Drugs Ther. 2023 Aug;37(4):729-741. doi: 10.1007/s10557-022-07331-1. Epub 2022 Apr 20. PMID 35441926
- [Background] Bernal-Jimenez MA, Calle G, Gutierrez Barrios A, Gheorghe LL, Cruz-Cobo C, Trujillo-Garrido N, Rodriguez-Martin A, Tur JA, Vazquez-Garcia R, Santi-Cano MJ. Effectiveness of an Interactive mHealth App (EVITE) in Improving Lifestyle After a Coronary Event: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2024 Apr 22;12:e48756. doi: 10.2196/48756. PMID 38648103
- [Background] Yilmaz E, Eser E, Sekuri C, Kultursay H. [The psychometric properties of the Turkish version of Myocardial Infarction Dimensional Assessment Scale (MIDAS)]. Anadolu Kardiyol Derg. 2011 Aug;11(5):386-401. doi: 10.5152/akd.2011.105. Epub 2011 Jun 7. Turkish. PMID 21652294
- [Background] Cruz-Cobo C, Bernal-Jimenez MA, Calle G, Gheorghe LL, Gutierrez-Barrios A, Canadas D, Tur JA, Vazquez-Garcia R, Santi-Cano MJ. Efficacy of a Mobile Health App (eMOTIVA) Regarding Compliance With Cardiac Rehabilitation Guidelines in Patients With Coronary Artery Disease: Randomized Controlled Clinical Trial. JMIR Mhealth Uhealth. 2024 Jul 25;12:e55421. doi: 10.2196/55421. PMID 39052330
- [Background] Turan Kavradim S, Canli Ozer Z. The effect of education and telephone follow-up intervention based on the Roy Adaptation Model after myocardial infarction: randomised controlled trial. Scand J Caring Sci. 2020 Mar;34(1):247-260. doi: 10.1111/scs.12793. Epub 2019 Nov 26. PMID 31769891
- [Background] Pietrzykowski L, Michalski P, Kosobucka A, Kasprzak M, Fabiszak T, Stolarek W, Siller-Matula JM, Kubica A. Medication adherence and its determinants in patients after myocardial infarction. Sci Rep. 2020 Jul 21;10(1):12028. doi: 10.1038/s41598-020-68915-1. PMID 32694522
- [Background] Varnfield M, Karunanithi M, Lee CK, Honeyman E, Arnold D, Ding H, Smith C, Walters DL. Smartphone-based home care model improved use of cardiac rehabilitation in postmyocardial infarction patients: results from a randomised controlled trial. Heart. 2014 Nov;100(22):1770-9. doi: 10.1136/heartjnl-2014-305783. Epub 2014 Jun 27. PMID 24973083
- [Background] Piepoli MF, Hoes AW, Agewall S, Albus C, Brotons C, Catapano AL, Cooney MT, Corra U, Cosyns B, Deaton C, Graham I, Hall MS, Hobbs FDR, Lochen ML, Lollgen H, Marques-Vidal P, Perk J, Prescott E, Redon J, Richter DJ, Sattar N, Smulders Y, Tiberi M, van der Worp HB, van Dis I, Verschuren WMM, Binno S; ESC Scientific Document Group. 2016 European Guidelines on cardiovascular disease prevention in clinical practice: The Sixth Joint Task Force of the European Society of Cardiology and Other Societies on Cardiovascular Disease Prevention in Clinical Practice (constituted by representatives of 10 societies and by invited experts)Developed with the special contribution of the European Association for Cardiovascular Prevention & Rehabilitation (EACPR). Eur Heart J. 2016 Aug 1;37(29):2315-2381. doi: 10.1093/eurheartj/ehw106. Epub 2016 May 23. No abstract available. PMID 27222591
- [Background] Gonzalez M, Sjolin I, Back M, Ogmundsdottir Michelsen H, Tanha T, Sandberg C, Schiopu A, Leosdottir M. Effect of a lifestyle-focused electronic patient support application for improving risk factor management, self-rated health, and prognosis in post-myocardial infarction patients: study protocol for a multi-center randomized controlled trial. Trials. 2019 Jan 24;20(1):76. doi: 10.1186/s13063-018-3118-1. PMID 30678709
- [Background] Ibanez B, James S, Agewall S, Antunes MJ, Bucciarelli-Ducci C, Bueno H, Caforio ALP, Crea F, Goudevenos JA, Halvorsen S, Hindricks G, Kastrati A, Lenzen MJ, Prescott E, Roffi M, Valgimigli M, Varenhorst C, Vranckx P, Widimsky P; ESC Scientific Document Group. 2017 ESC Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation: The Task Force for the management of acute myocardial infarction in patients presenting with ST-segment elevation of the European Society of Cardiology (ESC). Eur Heart J. 2018 Jan 7;39(2):119-177. doi: 10.1093/eurheartj/ehx393. No abstract available. PMID 28886621
- [Background] Johnston N, Bodegard J, Jerstrom S, Akesson J, Brorsson H, Alfredsson J, Albertsson PA, Karlsson JE, Varenhorst C. Effects of interactive patient smartphone support app on drug adherence and lifestyle changes in myocardial infarction patients: A randomized study. Am Heart J. 2016 Aug;178:85-94. doi: 10.1016/j.ahj.2016.05.005. Epub 2016 May 17. PMID 27502855
- [Background] Hançerlioğlu S, Aykar FŞ. Kronik Hastalıklarda Öz-Bakım Yönetimi Ölçeği'nin Türkçe'ye uyarlanması, geçerlik ve güvenirliği. GÜSBD. 2018;7:175-83
- [Background] Vrints C, Andreotti F, Koskinas KC, Rossello X, Adamo M, Ainslie J, Banning AP, Budaj A, Buechel RR, Chiariello GA, Chieffo A, Christodorescu RM, Deaton C, Doenst T, Jones HW, Kunadian V, Mehilli J, Milojevic M, Piek JJ, Pugliese F, Rubboli A, Semb AG, Senior R, Ten Berg JM, Van Belle E, Van Craenenbroeck EM, Vidal-Perez R, Winther S; ESC Scientific Document Group. 2024 ESC Guidelines for the management of chronic coronary syndromes. Eur Heart J. 2024 Sep 29;45(36):3415-3537. doi: 10.1093/eurheartj/ehae177. No abstract available. PMID 39210710
- [Background] Brown MT, Bussell JK. Medication adherence: WHO cares? Mayo Clin Proc. 2011 Apr;86(4):304-14. doi: 10.4065/mcp.2010.0575. Epub 2011 Mar 9. PMID 21389250
- [Background] Shang P, Liu GG, Zheng X, Ho PM, Hu S, Li J, Jiang Z, Li X, Bai X, Gao Y, Xing C, Wang Y, Normand SL, Krumholz HM. Association Between Medication Adherence and 1-Year Major Cardiovascular Adverse Events After Acute Myocardial Infarction in China. J Am Heart Assoc. 2019 May 7;8(9):e011793. doi: 10.1161/JAHA.118.011793. PMID 31057004
- [Background] Şen ET, Sertel Berk Ö, Sindel D. İlaç Uyumunu Bildirim Ölçeği'nin Türkçe uyarlamasının geçerlik ve güvenirlik çalışması. İstanbul Tıp Fakültesi Dergisi. 2019;82:52-61. doi: 10.26650/IUITFD.413637
- [Background] Ivers NM, Schwalm JD, Bouck Z, McCready T, Taljaard M, Grace SL, Cunningham J, Bosiak B, Presseau J, Witteman HO, Suskin N, Wijeysundera HC, Atzema C, Bhatia RS, Natarajan M, Grimshaw JM. Interventions supporting long term adherence and decreasing cardiovascular events after myocardial infarction (ISLAND): pragmatic randomised controlled trial. BMJ. 2020 Jun 10;369:m1731. doi: 10.1136/bmj.m1731. PMID 32522811
- [Background] Chow CK, Klimis H, Thiagalingam A, Redfern J, Hillis GS, Brieger D, Atherton J, Bhindi R, Chew DP, Collins N, Andrew Fitzpatrick M, Juergens C, Kangaharan N, Maiorana A, McGrady M, Poulter R, Shetty P, Waites J, Hamilton Craig C, Thompson P, Stepien S, Von Huben A, Rodgers A; TEXTMEDS Investigators*. Text Messages to Improve Medication Adherence and Secondary Prevention After Acute Coronary Syndrome: The TEXTMEDS Randomized Clinical Trial. Circulation. 2022 May 10;145(19):1443-1455. doi: 10.1161/CIRCULATIONAHA.121.056161. Epub 2022 May 9. PMID 35533220
- [Background] Du R, Wang P, Ma L, Larcher LM, Wang T, Chen C. Health-related quality of life and associated factors in patients with myocardial infarction after returning to work: a cross-sectional study. Health Qual Life Outcomes. 2020 Jun 17;18(1):190. doi: 10.1186/s12955-020-01447-4. PMID 32552846
- [Background] Salari N, Morddarvanjoghi F, Abdolmaleki A, Rasoulpoor S, Khaleghi AA, Hezarkhani LA, Shohaimi S, Mohammadi M. The global prevalence of myocardial infarction: a systematic review and meta-analysis. BMC Cardiovasc Disord. 2023 Apr 22;23(1):206. doi: 10.1186/s12872-023-03231-w. PMID 37087452
- [Background] Byrne RA, Rossello X, Coughlan JJ, Barbato E, Berry C, Chieffo A, Claeys MJ, Dan GA, Dweck MR, Galbraith M, Gilard M, Hinterbuchner L, Jankowska EA, Juni P, Kimura T, Kunadian V, Leosdottir M, Lorusso R, Pedretti RFE, Rigopoulos AG, Rubini Gimenez M, Thiele H, Vranckx P, Wassmann S, Wenger NK, Ibanez B; ESC Scientific Document Group. 2023 ESC Guidelines for the management of acute coronary syndromes. Eur Heart J. 2023 Oct 12;44(38):3720-3826. doi: 10.1093/eurheartj/ehad191. No abstract available. PMID 37622654
- See also: WHO. The top 10 causes of death — https://www.who.int/news-room/fact-sheets/detail/the-top-10-causes-of-death
- See also: WHO. Cardiovascular diseases (CVDs) — https://www.who.int/news-room/fact-sheets/detail/cardiovascular-diseases-(cvds)
- See also: WHO. Sodium reduction — https://www.who.int/news-room/fact-sheets/detail/salt-reduction
- See also: Hambraeus K, Hagström E, Leosdottir M. SEPHIA- Secondary prevention following coronary intensive care. SWEDEHEART Annual report 2016 — https://www.ucr.uu.se/swedeheart/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-02-05): https://cdn.clinicaltrials.gov/large-docs/44/NCT06882044/Prot_SAP_000.pdf